CLINICAL TRIAL: NCT01475942
Title: Randomized Placebo Controlled Study to Assess the Effect of a Probiotic Supplement on the Subclinical Levels of Intestinal C. Difficile Among Elderly
Brief Title: Probiotic Intervention With Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danisco (Industry)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Turku_elderly
Record Dates: First submitted 2011-09-20; First posted 2011-11-22 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-02

CONDITIONS: Intestinal C. Difficile
Keywords: elderly; probiotic; bowel function; pathogen; constipation; diarrhoea; Subclinical levels
MeSH Terms: conditions — Constipation; Diarrhea | interventions — Probiotics; Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Lactobacillus
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Sucrose
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — 4 month probiotic intervention with 1 month run-in and 1 month wash-out. Probiotic given once a day.
  Other Names: Lactobacillus

SUMMARY:
The study objective is to evaluate the effect of probiotic on faecal Clostridium difficile levels of elderly subjects.

DETAILED DESCRIPTION:
The study objective is to evaluate the effect of a probiotic Lactobacillus strain in lowering the levels of Clostridium difficile in the intestine of elderly subjects. In addition, the nutritional and general health status will be assessed using validated health related questionnaires. Bowel function and prevalence of infections will be followed throughout the intervention period. The study population consists of elderly home inhabitants. The study will be conducted as a double-blind placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* elderly subjects
* no acute infection at recruitment

Exclusion Criteria:

* antibiotic treatment 1 month prior to beginning of study
* less than 6 month life expectancy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in level of faecal Clostridium difficile | 0 weeks, 8 weeks, 16 weeks
  Quantification of C. difficile from faecal samples

SECONDARY OUTCOMES:
Change in nutritional status | 0 weeks, 16 weeks
  Evaluated according to the Mini Nutritional Assessment (MNA®) questionnaire.
Change in quality of life | 0 weeks, 16 weeks
  Evaluated according to the validated 15D© health related survey from adequately oriented subjects.
Change in levels of other intestinal pathogens than C. difficile | 0 weeks, 8 weeks, 16 weeks
  Quantified from faecal samples
Change in bowel function | 0 weeks, 16 weeks
  Assessed according to Bristol Stool Form Scale by health care personnel throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Sampo Lahtinen, PhD, Study Chair — Danisco; Anna Lyra, PhD, Study Director — Danisco; Matti Viitanen, MD, Principal Investigator — University of Turku
Locations (1):
- Elderly Home Kerttuli, Turku, Finland

IPD SHARING:
Plan to Share IPD: No